CLINICAL TRIAL: NCT05738278
Title: Heart Rate Informed Changes in Care for Non-Communicating Patients: A Randomized Controlled Trial
Brief Title: Heart Rate Informed Changes in Care for Non-Communicating Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Bjørnar Hassel, Professor, University of Oslo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: #2016/1956
Record Dates: First submitted 2022-10-27; First posted 2023-02-22 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder; Intellectual Disability; Communication, Nonverbal
Keywords: Heart Rate; Autistic Disorder; Intellectual Disability; Social Interaction; Caregivers; Developmental Disabilities; Communication; Biomarkers; Pain
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability; Nonverbal Communication; Autistic Disorder; Developmental Disabilities; Communication; Pain

STUDY DESIGN:
Intervention Model Description: Thirty-eight non-verbal patients are recruited. HR is taken as a marker of acute pain. HR-Variability (HRV) and pain-related inflammatory cytokines (MCP-1, IL-1RA, IL-8, TGFβ1, and IL-17) are collected as measures of long-term pain. Caregivers will be asked to what degree they observe pain in their patients and how well they believe they understand their patient's expression. Collection is set to primary care institutions. HR is measured 8 hours/day over 2 weeks to identify increase of HR associated with potentially painful situations. Changes in procedures are in the form of change in 1) rigorousness of stretching, 2) preparations for casts, 3) lifting technique, or 4) personal hygiene procedure. To differentiate effects due to procedure-change from effects of covariates such as increased attentiveness when using HR; half the study group will start intervention in week 3 while the delayed group will continue data collection for another 2 weeks before introducing procedure changes.
Who Masked: Outcomes Assessor
Masking Description: Due to the objectives of the study, the identity of test and control treatments will not be known when analysing data. Access to the randomization code will be strictly controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): After 2 weeks mapping phase, patient-specific HR-informed intervention from week 3.
  Interventions: Behavioral: HR-informed change in routine
- Control group (Active Comparator): After 4 weeks mapping phase, patient-specific HR-informed intervention from week 5.
  Interventions: Behavioral: Delayed HR-informed specific change in routine

INTERVENTIONS:
Behavioral: HR-informed change in routine — The intervention is given for a situation occuring at least ten times and accompanied by an increase in HR at least 80% of the time, during the two-week registration period. Change in care (intervention) is introduced from week 3.
  The intervention is in one of four forms:
  1. changes in physiotherapy, e.g., less rigorous movement in the identified painful stretch,
  2. preparations for putting on corrective cast to stabilize joint and/or stretch spastic muscles,
  3. change in procedures for transportation/lifting, e.g., new technique or adaptations made to equipment, or
  4. revised personal hygiene procedure.
  Arms: Intervention group
Behavioral: Delayed HR-informed specific change in routine — The intervention is given for a situation occuring at least twenty times and accompanied by an increase in HR at least 80% of the time, during the four-week registration period. Change in care (intervention) is introduced from week 5.
  The intervention is in one of four forms:
  1. changes in physiotherapy, e.g., less rigorous movement in the identified painful stretch,
  2. preparations for putting on corrective cast to stabilize joint and/or stretch spastic muscles,
  3. change in procedures for transportation/lifting, e.g., new technique or adaptations made to equipment, or
  4. revised personal hygiene procedure.
  Arms: Control group

SUMMARY:
The overarching aim is to generate knowledge to reduce incidence of pain in non-verbal patients' everyday life. The trial will 1) evaluate how HR can be used to identify potentially painful care procedures that should be re-evaluated in terms of the approach taken; 2) test the effect of heart rate (HR)-informed changes in potentially painful care procedures on biomarkers of pain, and 3) assess how six weeks of communication through HR affects the quality of communication between patient and caregiver.

DETAILED DESCRIPTION:
Detailed protocol to be published as journal article with reference to Clinicaltrials.gov-registration. Preprint available: https://osf.io/gan42

ELIGIBILITY:
Inclusion Criteria:

* Between 5 and 70 years of age at the time of data collection
* Autism spectrum disorder as evaluated by clinical psychologist
* Communication difficulties
* Living at a care home with round-the-clock staff for at least five days a week; or attending one-to-one staffed school/day-care at least five days a week.
* Written informed consent is obtained from the subjects' legal representative.

Exclusion Criteria:

- Having any autoimmune disorder or any type of cancer with ongoing chemotherapy.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Situations identified by 2 standard deviation increase in HR | 11 weeks
  The hypothesis is that a 2 standard deviation increase in HR can identify potentially painful care situations that require re-evaluation. Mean HR spike counts will be compared using a one-tailed paired sampled t-test to differentiate between suitable and unsuitable situations for care adjustments.

SECONDARY OUTCOMES:
HRV (ms) | 6 weeks
  The hypothesis is that HR-informed changes in a patient-specific care procedures will potentially painful settings and thus reduce pain-related biomarkers of HRV as evaluated at the beginning and the end of the study period.
Serum concentrations of MCP-1, IL-1RA, IL-8, TGFβ1, and IL-17 (pg/ml) | 6 weeks
  The hypothesis is that HR-informed changes in a patient-specific care procedures will potentially painful settings and thus reduce pain-related blood biomarkers (MCP-1, IL-1RA, IL-8, TGFβ1, and IL-17) as evaluated at the beginning and the end of the study period.
Scores on quality of communication | 6 weeks
  The hypothesis is that HR as an aid in communication will increase caregivers' understanding of the patient as measured by changes in perceived understanding of the patient from the beginning to the end of the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Bjørnar Hassel, Principal Investigator — University of Oslo
Locations (2):
- Norway (2):
  - Oslo University Hospital, Oslo
  - University of Oslo, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kildal E, Stadskleiv K, Boysen ES, Oderud T, Dahl IL, Seeberg TM, Guldal S, Strisland F, Morland C, Hassel B. Increased heart rate functions as a signal of acute distress in non-communicating persons with intellectual disability. Sci Rep. 2021 Mar 19;11(1):6479. doi: 10.1038/s41598-021-86023-6. PMID 33742078
- [Derived] Kildal ESM, Quintana DS, Szabo A, Tronstad C, Andreassen O, Naerland T, Hassel B. Heart rate monitoring to detect acute pain in non-verbal patients: a study protocol for a randomized controlled clinical trial. BMC Psychiatry. 2023 Apr 14;23(1):252. doi: 10.1186/s12888-023-04757-1. PMID 37060049